CLINICAL TRIAL: NCT00607464
Title: Multicentre Randomised Controlled Trial of HELP (Heat Loss Prevention) in the Delivery Room
Acronym: HeLP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Sunnybrook Health Sciences Centre (Other)
Collaborators: Canadian Institutes of Health Research (CIHR) (Other Government); Vermont Oxford Network (Network); University of Alberta (Other)
Responsible Party: Principal Investigator, Maureen Reilly, RRT, Sunnybrook Health Sciences Centre
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MCT-71137; ISRCTN85045728
Record Dates: First submitted 2008-01-22; First posted 2008-02-05 (Estimated); Last update posted 2016-04-25 (Estimated); Status verified 2016-04

CONDITIONS: Hypothermia in Premature Infants
Keywords: Hypothermia, premature infants, Polyethylene occlusive wrap
MeSH Terms: conditions — Hypothermia; Premature Birth

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Polyethylene occlusive skin wrap applied immediately after birth and removed after the infant has been admitted to a stable thermoneutral environment
  Interventions: Device: Polyethylene occlusive skin wrap
- 2 (No Intervention): Standard care

INTERVENTIONS:
Device: Polyethylene occlusive skin wrap — Polyethylene occlusive skin wrap applied immediately after birth and removed after the infant has been admitted to a stable thermoneutral environment
  Other Names: occlusive skin wrap
  Arms: 1

SUMMARY:
Does polyethylene occlusive wrap applied immediately after delivery to infants born at less than 28 weeks gestation decrease all-cause mortality measured at discharge compared with the standard of care as determined by the Neonatal Resuscitation Program guidelines (i.e. drying under radiant heat)?

DETAILED DESCRIPTION:
Thermoregulation is a major problem for low birth weight infants. The EPICure study showed that 36% of infants born between 24 and 25 weeks gestation had an admission temperature less than 35 degrees Celsius. Hypothermia is associated with increased risk of morbidity and mortality. The HeLP trial hopes to address these issues with the use of a polyethylene occlusive wrap applied immediately after delivery to infants born at less that 28 weeks gestation. Forty-five centers are currently involved in this study. Infant enrollments began in December 2004.

Primary outcome: To determine if polyethylene occlusive wrap applied immediately after delivery to infants born between 24+0 and 27+6 weeks gestation results in decreased mortality compared with the conventional method of drying. Because of increased mortality and variable center specific resuscitation practices, infants born at less than 24 weeks gestation will be randomized as part of a separate Pilot Study and centers may choose if they wish to participate in this group or not. Secondary outcome: The key secondary outcome will be axillary temperature taken on introduction into a warm environment in the NICU. We will also record clinically important variables including: acidosis, hypotension, hypoglycaemia, seizures, patent ductus arteriosus, respiratory distress syndrome/chronic lung disease, necrotizing enterocolitis and head ultrasound results. Length of stay and cause of death at discharge will also be recorded. Long-term follow-up is critical to our understanding of the implications of any new intervention. As such, we ask parents from hospitals who agree to participate in the follow-up study for permission to contact them approximately 18 months after birth.

Preterm infants meeting the eligibility criteria will be randomly assigned within three gestational age strata (less than 24 weeks, 24+0 to 25+6 weeks gestation, and 26+0 to 27+6 weeks gestation) to either the occlusive skin wrap group or the standard of care (non-wrap) group.

ELIGIBILITY:
Inclusion Criteria:Infants born at less than 28 weeks and who have prior to birth a firm decision to provide full resuscitative measures and intensive support.

-

Exclusion Criteria:1. Infants born with major congenital anomalies that are not covered by skin (e.g. gastroschisis, meningomyelocele) 2. Infants born with blistering skin conditions that preclude the use of occlusive wrap

-

Ages: 24 Weeks to 28 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 804 (Actual)
Dates: Start 2004-09; Primary Completion 2010-03 (Actual); Study Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Death to discharge or at six months corrected gestational age | discharge or six months corrected gestational age

SECONDARY OUTCOMES:
1. Axillary temperature upon arrival in Neonatal Intensive Care Unit (NICU) | upon arrival in NICU
acidosis, hypotension, hypoglycaemia, seizures | first 12 hours of life
4. Death and neurosensory disability measured at 18 months corrected gestational age | 18 months corrected gestational age
PDA, RDS, CLD, pneumothorax, sepsis, IVH, PVL, NEC, GI perforation, pulmonary hemorrhage, hearing, ROP | discharge from hospital or 6 months corrected gestational age

CONTACTS AND LOCATIONS:
Overall Officials: Maureen C Reilly, RRT, Principal Investigator — Sunnybrook Health Sciences Centre; Sunita Vohra, MD FRCPC MSc, Principal Investigator — University of Alberta/Stollery Children's Hospital
Locations (1):
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada

REFERENCES:
- [Derived] Reilly MC, Vohra S, Rac VE, Dunn M, Ferrelli K, Kiss A, Vincer M, Wimmer J, Zayack D, Soll RF; Vermont Oxford Network Heat Loss Prevention (HeLP) Trial Study Group. Randomized trial of occlusive wrap for heat loss prevention in preterm infants. J Pediatr. 2015 Feb;166(2):262-8.e2. doi: 10.1016/j.jpeds.2014.09.068. Epub 2014 Nov 12. PMID 25449224
- [Derived] Vohra S, Reilly M, Rac VE, Bhaloo Z, Zayack D, Wimmer J, Vincer M, Ferrelli K, Kiss A, Soll R, Dunn M. Study protocol for multicentre randomized controlled trial of HeLP (Heat Loss Prevention) in the delivery room. Contemp Clin Trials. 2013 Sep;36(1):54-60. doi: 10.1016/j.cct.2013.06.001. Epub 2013 Jun 11. PMID 23770234
- See also: The Vermont Oxford Network — http://www.vtoxford.org